CLINICAL TRIAL: NCT05713591
Title: Transition Care Model for Adolescents With Congenital Heart Disease (CHD): a Multicenter Study to Assess Its Effectiveness on Patient-reported Outcomes (TELEMACO Study)
Brief Title: Transition Care Model for Adolescents With Congenital Heart Disease
Acronym: TELEMACO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Serena Francesca Flocco, Principal Investigator, IRCCS Policlinico S. Donato
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Supportive Care
Other Study IDs: 127/int/2019
Record Dates: First submitted 2023-01-25; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Congenital Heart Disease
Keywords: congenital heart disease; transition care; quality of life; engagement
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: The model of Transition Care (TC) is a complex educational intervention that encompasses three main steps (first step: understanding of their clinical condition; second step: education and support; third step: involvement and collaboration). Each step was developed to include, simplify and standardize the implementation of targeted and personalized interventions.
  After the eligibility criteria check, patients will be randomized in experimental or control arms. Patients in the experimental arm were involved in the model TC, while patients in the control group received the standard of care. Data collection for each group was performed at baseline and at three, six, nine, and twelve months.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Eligible patients who signed the written informed consent will be blindly randomized (allocation 1:1) in each involved CHD center at the baseline phase. However, considering the type of interventions is not possible to guarantee the patients' blindness during the study, as well as for the care provider.
  The eligible patients will be randomized by using a pre-determined randomization sheet that considers patients' entry ID (the chronological number of enrollment) to perform randomization (each CHD center that participates in the research project will have a specific pre-determined randomization sheet). Patients will be randomized on a 1:1 basis to receive the TC model or usual care during the transition from childhood to adulthood.
  Only the outcome assessor and the principal investigator will be blind to the patient allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transition care model (Experimental): Patients in the experimental arm will receive the TC intervention which encompasses three main pillars that guided a standardized and structured clinical pathway to ensure an optimal transition from childhood care to adult care. Briefly, the first pillar was designed to improve the understanding of the clinical condition through tailored education. Healthcare providers delivered specific information and education strategies. The second pillar aimed to support the development of functional coping strategies by discussing with a counselor and/or a psychologist. The TC encompassed for this pillar both structured face-to-face discussions and counseling moments. The third pillar hoped to improve the engagement of CHD adolescents and their families.
  Interventions: Behavioral: Transition care model
- Usual care (No Intervention): Patients in the control arm will receive a usual care approach without the high focus on standardization given by the experimental arm (e.g. without flyers and booklets or standardized moments of face-to-face counseling). Data collection will be performed using a consistent approach with the one described in the experimental arm: every three months in a year (T0, T1, T2, T3, and T4).

INTERVENTIONS:
Behavioral: Transition care model — The transition care model (TC) consists in multidisciplinary standardized interventions to educate and support adolescents with congenital heart disease, representing a key element in the adequate delivery of care to these individuals during their transition from childhood to adulthood. This model encompasses three main pillars previously described.
  Arms: Transition care model

SUMMARY:
The primary aim of this study is to assess the effectiveness of a standardized transition care model (TC) on the perceived mental and physical health of adolescents with congenital heart disease (CHD). Furthermore, the secondary aims of this research are focused on providing a description of the impact of a standardized TC on overall healthcare needs, satisfaction, and engagement.

Therefore, a prospective, randomized, controlled, single-blind, and multi-center study will be conducted.

DETAILED DESCRIPTION:
Congenital heart diseases (CHD) are some of the most prevalent and serious birth defects, representing a major global health problem. With a prevalence of 9.1 for 1000 live births, the CHD are the leading causes of birth defects associated with morbidity, mortality, and medical expenditures. Currently, 1.3 million children live with a CHD worldwide (3), and approximately 90% of them can survive into adulthood. In this scenario, the transition from childhood to adulthood is one of the most complex and delicate part of life for CHD patients. The multi-disciplinary standardized interventions to educate and support patients with CHD, described as "Transition Clinic" (TC), represent a key element in delivering care for patients during the transition from childhood to adulthood. However, most recent literature focuses on the CHD childhood clinical management or the CHD adulthood challenges (i.e., GUCH challenges). Thus, the attention to exploring the peculiarities of the transition period from childhood to adulthood in patients with CHD is underinvestigated by the lack of experimental studies [i.e. randomized controlled trial (RCT)] as the published evidence is related to the assessment of effects of the same model on outcomes without a control arm (pre-post test study design).

ELIGIBILITY:
Inclusion Criteria:

* Adolescent patients (aged between 12 and 18 years)
* Diagnosis of CHD, according to 2018 AHA/ACC Guideline for the Management of Adults With Congenital Heart Disease
* All patients who express the willingness to participate in the study through the signing of the informed consent form and signature of informed consent by patients' parents
* Moderate and Complex CHD, according to the classification described by Warnes

Exclusion Criteria:

* Chromosomal abnormalities such as Down's syndrome and Marfan's syndrome
* Patients with cognitive impairment (assessed using Six Item Screener, SIS): if SIS ≤4
* Not understanding the Italian language
* Patients in pregnancy
* Simple CHD, according to Warnes (2001) (25).

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 964 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical and mental quality of life | up to 12 months
  This outcome will be measured through a self-report tool such as a short-form survey. The short-form survey allows for assessing physical and mental health. The score will be computed for each domain and a higher score indicates a better perception of quality of life.

SECONDARY OUTCOMES:
Engagement | Every 3 months from baseline, up to 12 months
  Patient engagement will be measured through the Patient Health Engagement scale. The score will be computed based on four main constructs: blackout, arousal, adhesion, and eudaimonic project. The final score has been computed through the median of the values of each item, ranging from 1 to 7, and a higher score indicates a better perception of engagement.
Healthcare needs | Every 3 months from baseline, up to 12 months
  Adolescent healthcare needs will be measured through the Healthcare Needs Scale for Youth with congenital heart disease during the transition to adulthood. The score will be computed based on four main constructs: healthcare education, clinical support, emotional support, and continuum of care. The final score ranged from 0 to 100 and higher scores indicate higher needs.
Satisfaction of patients | Every 3 months from baseline, up to 12 months
  Adolescent satisfaction will be measured through the visual analog scale. The VAS consists of a 10 cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, MI, Italy

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.